CLINICAL TRIAL: NCT06828627
Title: Laparoscopic Total Left-sided Surgical Approach Versus Traditional Bilateral Surgical Approach for Treating Hiatal Hernia: a Randomized Controlled Trial
Brief Title: Laparoscopic Total Left-sided Surgical Approach Versus Traditional Bilateral Surgical Approach for Hiatal Hernia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ChiCTR2000034028
Record Dates: First submitted 2025-01-21; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2020-07

CONDITIONS: Hiatal Hernia; GERD
Keywords: surgical approach; efficacy; safety; randomized controlled trial
MeSH Terms: conditions — Hernia, Hiatal; Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Total left-sided surgical approach; TLSA (Experimental): TLSA surgery procedure. (A) On the greater curvature of the stomach, the gastrocolic ligament is incised along the avascular area between the left and right gastric omentum vessels, and the gastric fundus is separated upward to the cardia to protect the vagus nerve.
  (B) The cardia, lower esophagus, and diaphragm is exposed, and the confluence of the left and right crus of the diaphragm is revealed.
  The retroperitoneum at the left and right crus of the diaphragm is incised, and the lower esophagus is dissociated for about 3-5 cm. The gastric fundus and the posterior wall of the esophagus are fully dissociated from the upper spleen. (C) Non-absorbable thread is used to intermittently suture the left and right crus of diaphragm in order to reconstruct the esophagus hiatus with a diameter of about 1.5 cm. (D) Then, the surgeon inserts the patch and fixes it on the crus of diaphragm if the hiatal hernia is larger than 5 cm or the diaphragm on both sides is weak. (E) A small incision
  Interventions: Procedure: TLSA
- Traditional bilateral surgical approach; TBSA (Active Comparator): Traditional bilateral surgical approach (TBSA) surgery procedure. (A) Separation is initiated from the avascular area of the lesser omentum, and the hepatic branch of vagus nerve is preserved as far as possible. Careful separation is performed upward to expose the right crus of diaphragm. (B) At the greater curvature of the stomach, two to three short gastric vessels are cut off to expose the left crus of diaphragm, and the space between the anterior and posterior of esophagus is dissociated. (C) The diaphragmatic esophageal membrane is incised and the lower part of the esophagus is dissociated about 4-5 cm, then the gastroesophageal valve flap is reformed and the His angle is restored. During the operation, it mainly protects the anterior and posterior trunk of the vagus nerve. The anterior and posterior trunk of the vagus nerve are mainly protected during the operation. (D) Both sides of the crus of the diaphragm are intermittently sutured with non-absorbable thread to recons
  Interventions: Procedure: TBSA

INTERVENTIONS:
Procedure: TLSA — TLSA surgery procedure. (A) On the greater curvature of the stomach, the gastrocolic ligament is incised along the avascular area between the left and right gastric omentum vessels, and the gastric fundus is separated upward to the cardia to protect the vagus nerve.
  (B) The cardia, lower esophagus, and diaphragm is exposed, and the confluence of the left and right crus of the diaphragm is revealed.
  The retroperitoneum at the left and right crus of the diaphragm is incised, and the lower esophagus is dissociated for about 3-5 cm. The gastric fundus and the posterior wall of the esophagus are fully dissociated from the upper spleen. (C) Non-absorbable thread is used to intermittently suture the left and right crus of diaphragm in order to reconstruct the esophagus hiatus with a diameter of about 1.5 cm. (D) Then, the surgeon inserts the patch and fixes it on the crus of diaphragm if the hiatal hernia is larger than 5 cm or the diaphragm on both sides is weak. (E) A small incisio
  Arms: Total left-sided surgical approach; TLSA
Procedure: TBSA — Traditional bilateral surgical approach (TBSA) surgery procedure. (A) Separation is initiated from the avascular area of the lesser omentum, and the hepatic branch of vagus nerve is preserved as far as possible. Careful separation is performed upward to expose the right crus of diaphragm. (B) At the greater curvature of the stomach, two to three short gastric vessels are cut off to expose the left crus of diaphragm, and the space between the anterior and posterior of esophagus is dissociated. (C) The diaphragmatic esophageal membrane is incised and the lower part of the esophagus is dissociated about 4-5 cm, then the gastroesophageal valve flap is reformed and the His angle is restored. During the operation, it mainly protects the anterior and posterior trunk of the vagus nerve. The anterior and posterior trunk of the vagus nerve are mainly protected during the operation. (D) Both sides of the crus of the diaphragm are intermittently sutured with non-absorbable thread to reconst
  Arms: Traditional bilateral surgical approach; TBSA

SUMMARY:
Background: In China, guidelines for the treatment of hiatal hernia (HH) are lacking. Furthermore, efficacy and safety assessments of surgical approaches for HH and for the protection of the vagus nerve and organ function are needed. Therefore, the present clinical trial is being conducted to establish the normative treatment for HH. Methods: The current trial is an ongoing, single-center, randomized controlled trial of patients with HH. The total sample size required for the trial (July 2020-December 2023) is approximately 114 patients.

Patients will be randomly assigned to either an experimental group (total left-sided surgical approach; TLSA) or a control group (traditional bilateral surgical approach; TBSA) at a ratio of 1:1 using the block randomization method. We will use case report forms (CRFs) and electronic data capture (EDC) systems to obtain demographic information, preoperative laboratory tests, auxiliary examination results, operation information, and postoperative condition. The patients will be followed up for 3 years after surgery. The primary endpoint is the gastrointestinal quality-of-life index (GIQLI) at 1 year. The secondary endpoints include an efficacy evaluation index [consisting of the incidence of gallstones and gastric emptying disorders, gastrointestinal function recovery time, visual analog scale (VAS) scores, objective evaluation of postoperative indices, and surgical information] and a safety evaluation index (consisting of the incidence of postoperative complications, the 30-day postoperative mortality rate, and the HH recurrence rate at 1 and 3 years after surgery). Discussion: TLSA can protect the normal physiological function of organs to a certain extent by protecting the vagus nerve from injury, and has satisfactory short- and long-term efficacy. There is no significant difference in the incidence of postoperative complications and surgical safety between TLSA and TBSA. Our findings will facilitate clinical decision-making for HH and improve the life quality of patients.

Trial registration: Chinese Clinical Trial Registry, ChiCTR2000034028 (registration date: June 21, 2020). Keywords: Hiatal hernia (HH); surgical approach; efficacy; safety; randomized controlled trial

ELIGIBILITY:
Inclusion Criteria:

* (I) HH (type II/III/IV) diagnosed by gastroscopy, high-resolution esophageal manometry, and 24-hour esophageal pH monitoring.

(II) Aged 18-65 years, with no sex restrictions. (III) Eastern Cooperative Oncology Group score of ≤2 points and an American Society of Anesthesiologists score of ≤2 points.

Exclusion Criteria:

- (I) patients with cerebrovascular injury that occurred within the 6 months prior, unstable angina, or myocardial infarction; (II) patients with a history of uncontrolled epilepsy, central nervous system disease, or malignant tumor, or those with impaired judgment or mental illness who cannot cooperate with the research (III) patients with a history of digestive system tumors, or thoracic or abdominal surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
gastrointestinal quality-of-life index (GIQLI) | postoperative 1-year
  GIQLI is related to the QOL for gastrointestinal disorders. It contains 5 subscales, with a total score of 144 points. The higher the score, the better the patient's QOL and the better the surgical effect.
esophagitis | 3 years after surgery
  varified by gastroscopy （LA-standard）
DeMeester score | 3 years after surgery
  varified by high-resolution esophageal manometry and 24-hour esophageal pH monitoring； >4% indicate abnormal acid reflux

SECONDARY OUTCOMES:
Incidence of gallstones | postoperative 3-year
Incidence of gastric emptying disorders | 1 year after surgery
gastrointestinal function recovery time | 3 years after surgery
blood glucose | 3 years after surgery
serum lipid levels | 3 years after surgery
operation time | From enrollment to the end of treatment
blood loss | From enrollment to the end of treatment
abdominal drainage fluid volume, | From treatment to 30-days after surgery
total duration of hospitalization | From treatment to 30-days after surgery
incidence of postoperative complications | From treatment to 30-days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes